CLINICAL TRIAL: NCT03641742
Title: The Families-At-risk for Interstitial Lung Disease Study
Brief Title: Families-At-risk for Interstitial Lung Disease Study
Acronym: FAR-ILD
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: University of Washington (Other); Weill Medical College of Cornell University (Other); University of Iowa (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christine Garcia, Frode Jensen Professor of Medicine, Columbia University
Other Study IDs: AAAR1916; 2R01HL103676-05 (NIH)
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
Keywords: Interstitial Lung Disease; Pulmonary Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Tissue samples
  * Airway Brushings
  * Urine
  * Bronchoalveolar Lavage Fluid
  * Buccal swab and or saliva; only if blood is unavailable.
  * Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FAR-ILD Proband Participants: There will be no interventions administered to this group, only data collection.
- FAR-ILD "At-Risk" Participants: There will be no interventions administered to this group, only data collection

SUMMARY:
The interstitial lung diseases (ILDs) are a family of closely related lung conditions characterized by alveolar inflammation, injury, and fibrosis not due to infection or neoplasia. While previously considered to be rare, a recent nationwide study found that idiopathic pulmonary fibrosis (IPF), a fibrotic ILD with a median survival of only 3.8 years, affects nearly 0.5% of older adults in the U.S. While pirfenidone and nintedanib slow the progression of IPF, neither reverses fibrosis nor prevents progression of the disease,and no studies to date have tested interventions that prevent the development of fibrotic ILDs.

DETAILED DESCRIPTION:
The NHLBI has prioritized research focused on the primary prevention of chronic lung diseases, including ILD. The overall goal of this study is to conduct studies preparatory to and requisite for the testing of ILD preventative interventions.

In the current study, the investigators propose to examine the pulmonary histopathology and biology of early subclinical ILD in healthy adults with a first-degree relative with clinically diagnosed ILD. There are two currently accepted computed tomographic (CT)-based phenotypes of subclinical ILD: high attenuation areas (HAAs) and interstitial lung abnormalities (ILA). Investigators from Columbia University Medical Center have previously shown that HAA has strong construct validity as an imaging biomarker of early subclinical alveolar inflammation and fibrosis among community-dwelling adults using the Multi-Ethnic Study of Atherosclerosis (MESA), an ongoing NHLBI-funded prospective cohort study of 6,814 adults age 45 and older at enrollment in 2000-02. Investigators found that greater HAA at baseline was independently associated with reduced lung function and exercise capacity at 5-year follow-up, exertional dyspnea at 10-year follow-up, and elevated serum levels of matrix metalloproteinase-7 (MMP-7) and interleukin-6 (IL-6). ILA is a distinct qualitative and visually-identified early ILD phenotype on CT that has also shown strong construct validity for ILD. Neither HAA nor ILA has been validated histopathologically.

The lipoprotein substudy will examine the role of high density lipoproteins in patients with ILD. Patients with IPF have previously been shown to have low levels of high density lipoprotein (HDL) and high levels of low density lipoprotein (LDL). Investigators have previously shown that high levels of high-density cholesterol (HDL-C) are associated with a reduction in lung injury, inflammation and fibrosis (subclinical ILD) on CT in community-dwelling adults enrolled in the Multi-Ethnic Study of Atherosclerosis. These data are consistent with animal model data showing that treatment with apolipoprotein A-I (ApoA-I; the main component of HDL) attenuates lung fibrosis. Investigators at Columbia University Medical Center are therefore proposing to examine the associations of HDL and its main components (apolipoprotein A-I, apolipoprotein A-II, and paraoxonase-1) with clinical outcomes (FVC decline, death, lung transplantation and respiratory hospitalizations) and serum biomarkers of lung injury, inflammation and remodeling (SP-A, MMP-7, ICAM-1, IL-1, IL-18) in patients with ILD. Investigators will also explore the structure (using quantitative proteomics) and function (using a macrophage efflux assay and paraoxonase-1 activity assay) of HDL particles in adults with ILD and first-degree family members with subclinical ILD.

Obstructive sleep apnea (OSA) is highly prevalent among adults with interstitial lung disease (ILD) and maybe a risk factor based on our previous studies from MESA (https://www.mesa-nhlbi.org/) and other research studies completed at Columbia University Medical Center. Therefore, the investigators will examine the association between OSA and sub-clinical ILD in at-risk adults.

ELIGIBILITY:
Inclusion Criteria: For "At Risk" participants without clinical ILD

* Age 35 years or older, however subjects who are 40 years old and above will undergo HRCT and subjects age 40-65 years old will be eligible to undergo bronchoscopy
* First-degree relative with one of the following clinical diagnoses:
* Idiopathic Pulmonary Fibrosis
* Idiopathic Non-Specific Interstitial Lung Disease (with fibrosis)
* Chronic Hypersensitivity Pneumonitis (with fibrosis)
* Unclassifiable Idiopathic Interstitial Pneumonia (with fibrosis)
* Patients with any ILD characterized by fibrosis on CT chest scan
* Ability to provide informed consent

Inclusion Criteria: For "At Risk Smoker" participants without clinical ILD

* At least 50 years of age
* Smoked at least 1 pack a day for 30 years

Exclusion Criteria: For "At-Risk" participants without clinical ILD

* Known history of interstitial lung disease
* History of illicit drug use within the past year.
* Lower respiratory tract infection in the past 90 days.
* History of chest CT scan in the past year.
* Known history of heart failure or chronic kidney or liver disease.
* Pregnancy or Lactation

Inclusion Criteria: For "Proband" participants with clinical ILD Age 18 years or older

* Has one of the following clinical diagnoses as per ATS guidelines:
* Idiopathic Pulmonary Fibrosis
* Idiopathic Non-Specific Interstitial Lung Disease (with fibrosis)
* Chronic Hypersensitivity Pneumonitis (with fibrosis)
* Unclassifiable Idiopathic Interstitial Pneumonia (with fibrosis)
* Patient with any ILD characterized by fibrosis on CT chest scan
* Ability to provide informed consent

Exclusion Criteria: For "Proband" participants with clinical ILD

* No Living 1st degree relatives.

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants with and without a diagnosis of Interstitial Lung Disease. Adult participants with a diagnosis of interstitial lung disease as per American Thoracic Society (ATS) guidelines. Adult participants with a first-degree relative with a clinical diagnosis of interstitial lung disease. Adult participants who are at least 50 years of age with a smoking history of a minimum of 1 pack per day.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Garcia, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will be required to submit a written request to the PI describing the use of the data. The researcher must also document institutional review board (IRB) approval. No identifiable information will be released.
Access Criteria: De-identified data.

REFERENCES:
- [Background] Ost DE, Ernst A, Lei X, Kovitz KL, Benzaquen S, Diaz-Mendoza J, Greenhill S, Toth J, Feller-Kopman D, Puchalski J, Baram D, Karunakara R, Jimenez CA, Filner JJ, Morice RC, Eapen GA, Michaud GC, Estrada-Y-Martin RM, Rafeq S, Grosu HB, Ray C, Gilbert CR, Yarmus LB, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic Yield and Complications of Bronchoscopy for Peripheral Lung Lesions. Results of the AQuIRE Registry. Am J Respir Crit Care Med. 2016 Jan 1;193(1):68-77. doi: 10.1164/rccm.201507-1332OC. PMID 26367186
- [Background] Facciolongo N, Patelli M, Gasparini S, Lazzari Agli L, Salio M, Simonassi C, Del Prato B, Zanoni P. Incidence of complications in bronchoscopy. Multicentre prospective study of 20,986 bronchoscopies. Monaldi Arch Chest Dis. 2009 Mar;71(1):8-14. doi: 10.4081/monaldi.2009.370. PMID 19522159
- [Background] Pue CA, Pacht ER. Complications of fiberoptic bronchoscopy at a university hospital. Chest. 1995 Feb;107(2):430-2. doi: 10.1378/chest.107.2.430. PMID 7842773
- [Background] Jin F, Mu D, Chu D, Fu E, Xie Y, Liu T. Severe complications of bronchoscopy. Respiration. 2008;76(4):429-33. doi: 10.1159/000151656. Epub 2008 Aug 21. PMID 18716395
- [Background] Rosenthal E. New York seeks to tighten rules on medical research. N Y Times Web. 1996 Sep 27:B4. No abstract available. PMID 11648036

RESULTS

PARTICIPANT FLOW:
Groups:
- FAR-ILD Proband Participants: Historic data (from medical records) were reviewed.
- FAR-ILD "At-Risk" Participants: Individuals underwent CT chest imaging and Pulmonary Function testing.
Period: Overall Study
Arm/Group | FAR-ILD Proband Participants | FAR-ILD "At-Risk" Participants
Started | 27 | 98
Completed | 27 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAR-ILD Proband Participants | FAR-ILD "At-Risk" Participants | Total
Number analyzed (Participants) | 27 | 98 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 89 | 96
  >=65 years | 20 | 9 | 29
Age, Continuous [Mean (Full Range); unit: years] — Age at the time of enrollment, in years
  years | 68 [29 to 87] | 52 [37 to 77] | 54 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 61 | 71
  Male | 17 | 37 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only 18 of 57 probands signed consent forms; their data is included here.
  Participants
    Hispanic or Latino | 5 | 25 | 30
    Not Hispanic or Latino | 22 | 73 | 95
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 22 | 72 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 21 | 24
Region of Enrollment [Number; unit: participants]
  United States | 27 | 98 | 125
Interstitial Lung Abnormality (ILA) [Count of Participants; unit: Participants] — Computed tomography imaging of the chest that shows abnormalities of the lung parenchyma
  Participants | 27 | 0 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ILA (Interstitial Lung Abnormalities)
Description: The visual identification of the presence of ILA (Interstitial Lung Abnormalities) on CT chest scan by a thoracic radiologist.
Time Frame: During imaging (up to 1 hour)
Measure: Count of Participants; unit: Participants
Groups:
- FAR-ILD "At Risk" Participants Without ILA: The number of "At Risk" Participants whose Chest CT imaging, which was obtained as part of this study, did not show Interstitial Lung Abnormalities (ILA)
- FAR-ILD "At-Risk" Participants With ILA: The number of "At Risk" Participants whose CT imaging, which was obtained as part of this study, showed evidence of Interstitial Lung Abnormalities (ILA)
Arm/Group | FAR-ILD "At Risk" Participants Without ILA | FAR-ILD "At-Risk" Participants With ILA
Number analyzed (Participants) | 98 | 98
Participants | 85 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data collected through study completion, an average of 1 year.
Groups:
- FAR-ILD Proband With an Adverse Event; FAR-ILD "At-Risk" Participant With and Adverse Event: Any adverse event resulting from participation in the study.
Arm/Group | FAR-ILD Proband With an Adverse Event | FAR-ILD "At-Risk" Participant With and Adverse Event
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/98
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/98
Other Adverse Events (participants affected / at risk) | 0/27 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAR-ILD Proband With an Adverse Event (N=27) | FAR-ILD "At-Risk" Participant With and Adverse Event (N=98)
Death due to respiratory cause (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient died from progressive pulmonary fibrosis and advanced disease during the time frame of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03641742/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT03641742/ICF_001.pdf